CLINICAL TRIAL: NCT06946784
Title: LIFE-TB ; Long-Term Impacts on Lung Health and Life After Tuberculosis in Korea
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-1620
Record Dates: First submitted 2025-04-13; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis; Post Tuberculosis
Keywords: post tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active TB patients initiating or undergoing treatment or Post-treatment TB survivors

SUMMARY:
This is a prospective, multicenter observational cohort study aimed at establishing a nationwide post-TB lung disease registry in Korea. The study will enroll adult participants either undergoing treatment for pulmonary tuberculosis or with a history of treated TB. Over a five-year follow-up period, the study will assess the long-term health consequences of TB, focusing on respiratory symptoms, radiological changes, pulmonary function, and quality of life.

DETAILED DESCRIPTION:
"The LIFE-TB (Long-Term Impacts on Lung Health and Life After Tuberculosis in Korea) study is a nationwide, prospective, multicenter observational cohort designed to systematically investigate the long-term impacts of tuberculosis (TB) on lung health and quality of life. This registry aims to fill the critical evidence gap in understanding post-TB lung disease (PTLD) by enrolling adults with a current diagnosis of pulmonary TB or a history of TB treatment.

Participants will be recruited from six tertiary care centers across Korea. Eligible individuals include those aged 19 or older who are either undergoing anti-TB treatment or have completed it. Exclusion criteria include extrapulmonary TB without lung involvement, age under 19, or refusal to consent.

Data will be collected at baseline and regularly over a five-year follow-up period. Clinical variables include demographic information (age, sex, BMI, smoking status), TB-related history (sputum smear/culture, drug resistance, treatment outcomes), comorbidities, and current medications. Clinical assessments involve standardized symptom scores (mMRC), chest imaging (X-ray and CT), spirometry, and validated instruments to assess quality of life (EQ-5D-5L, PROMIS, SGRQ). Laboratory data include blood tests (HbA1c, lipids), HIV/HBV/HCV status, and urine and ECG assessments at baseline.

Participants will be followed annually, with interim assessments including imaging, spirometry, and symptom scoring at specified intervals. No study-specific interventions or additional imaging are required beyond routine care. Chest CTs will only be collected if obtained for clinical purposes.

The study's primary objectives are to describe the prevalence and trajectory of PTLD-related abnormalities and identify factors associated with poor outcomes. Secondary analyses include trends in pulmonary function and quality of life over time, as well as health utilization patterns. Statistical analyses include descriptive statistics and multivariable logistic regression to identify risk factors.

All data will be anonymized and securely stored, following institutional and ethical guidelines. The study will contribute essential real-world data to inform national and international post-TB management strategies."

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years
* Diagnosed with pulmonary TB and either initiating or undergoing treatment or history of treated pulmonary TB

Exclusion Criteria:

* Age <19 years
* Extrapulmonary TB without lung involvement
* Refusal to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants either undergoing treatment for pulmonary tuberculosis or with a history of treated TB.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
respiratory symptoms | 6month , 1year, 2year, 3year, 4year, 5year, 6year
  Prevalence and progression of respiratory symptoms (mMRC score, cough, sputum, hemoptysis)
abnormal radiographic findings | 6month , 1year, 2year, 3year, 4year, 5year, 6year
  abnormal findings of chest X-ray or chest CT
pulmonary function | 6month , 1year, 2year, 3year, 4year, 5year, 6year
  Pulmonary function measured by spirometry: FEV1, FVC, FEV1/FVC
Quality of life | 6month , 1year, 2year, 3year, 4year, 5year, 6year
  Quality of life measured by EQ-5D-5L, PROMIS, SGRQ

SECONDARY OUTCOMES:
poor long-term outcome | 6month , 1year, 2year, 3year, 4year, 5year, 6year
  Association of poor long-term outcomes with demographic and clinical variables (age, sex, BMI, comorbidities)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine Division of Pulmonology, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung C, Min J, Jeon D, Kwon YS, Mok J, Kim HW, Park Y, Kang YA. Protocol of a Nationwide Observational Cohort Study for Long-Term Impacts on Lung Health and Life after Tuberculosis in Korea (LIFE-TB). Tuberc Respir Dis (Seoul). 2026 Jan;89(1):86-93. doi: 10.4046/trd.2025.0109. Epub 2025 Oct 15. PMID 41088970